CLINICAL TRIAL: NCT00765557
Title: Randomized, Double-Blinded, Placebo-Controlled Trial of Laxatives for Children With Urge Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Department of Urology (Unknown)
Responsible Party: Principal Investigator, Linda A Baker, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: STU 122004-038
Record Dates: First submitted 2008-09-30; First posted 2008-10-03 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Constipation
Keywords: Bowel and bladder dysfunction; Constipation; MiraLAX; Overactive bladder; Polyethylene glycol; Urinary urgency
MeSH Terms: conditions — Constipation; Urinary Bladder, Overactive | interventions — polyethylene glycol 3350; Polyethylene Glycols; Glucose

STUDY DESIGN:
Intervention Model Description: A prospective randomized, double-blind, placebo controlled study was performed to determine whether placebo-controlled versus Polyethylene glycol (MiraLAX) was effective for decreasing OAB symptoms.
Who Masked: Participant, Investigator
Masking Description: The Investigational Drug Pharmacist will be blinded to all patient data, and physicians and nurses evaluating patients will be blinded to randomization of these patients to laxative versus placebo arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MiraLAX (Active Comparator): The Investigational Drug Pharmacist will be blinded to all patient data, and physicians and nurses evaluating patients will be blinded to randomization of these patients to MiraLAX versus placebo.
  Interventions: Drug: MiraLAX; Drug: Placebos
- Placebos (Placebo Comparator): The Investigational Drug Pharmacist will be blinded to all patient data, and physicians and nurses evaluating patients will be blinded to randomization of these patients to placebo versus MiraLAX.
  Interventions: Drug: MiraLAX; Drug: Placebos

INTERVENTIONS:
Drug: MiraLAX — Every subject will be given one bottle of the polyethylene glycol/placebo, divided into daily doses and depending on the patient's age, will be instructed to take 8.5 grams or 17 grams of the medication dispensed in daily dose vials to be mixed with water or juice. They will take the medication once a day for one month.
  Other Names: Polyethylene glycol
Drug: Placebos — Every subject will be given one bottle of the polyethylene glycol/placebo, divided into daily doses and depending on the patient's age, will be instructed to take 8.5 grams or 17 grams of the medication dispensed in daily dose vials to be mixed with water or juice. They will take the medication once a day for one month.
  Other Names: Dextrose

SUMMARY:
HYPOTHESIS:

Is MiraLAX an effective treatment of pediatric urinary urge syndrome?

OBJECTIVE:

Polyethylene glycol (PEG) is common first-line therapy for urinary symptoms despite minimal evidence-based support. We performed a randomized, double-blind, placebo-controlled study of PEG for initial treatment of urinary urge symptoms.

SUMMARY:

Only patients of investigators and sub-investigators will be recruited for this study. Children with urinary incontinence, urinary frequency, diurnal incontinence, Urinary Tract Infection (UTI) and/or reflux validated by bladder/bowel symptom questionnaire to have Urge Syndrome (US) are eligible for this study. A standardized questionnaire of bowel/bladder activity will be administered and a KUB obtained as standard of care at entry to the study. A standard 1-day voiding diary will be completed at home before beginning therapy. To exclude patients potentially still in the process of toilet training, only subjects 4 years of age and older will be studied. Other exclusion criteria will include known neurological disorders, a diagnosis of attention deficit disorder, bladder symptoms less than 6 months in duration at presentation, other bladder dysfunctions besides US, a history of anorectal malformation and pregnancy. Based upon prior experience that patients with encopresis were not likely to achieve improved stooling with only a few weeks of laxative therapy, they will also be excluded.

Those accepted into the study will be randomized to receive either laxative or placebo once daily for one month. Preparation of the laxative and placebo and patient randomization will be performed by the Children's Medical Center Investigational Drug Pharmacist. Premixed study medications will be available at the Urology clinic ready to be dispensed to the patient by the study coordinator after being screened and randomized. Dosage includes children age 4-6 years (8.5 gms) and children 7-10 years (17gms). The medication will be divided into daily doses by the Investigational Pharmacist. Written and verbal instructions, both in English and Spanish, will be provided to the parents/guardian of the subjects.

The Investigational Drug Pharmacist will be blinded to all patient data, and physicians and nurses evaluating patients will be blinded to randomization of these patients to laxative versus placebo arms.

DETAILED DESCRIPTION:
Urge Syndrome (US) is the most common non-neurogenic voiding dysfunction in children beyond the usual age for toilet training, and is characterized by urinary frequency and urgency, holding maneuvers, and diurnal incontinence. Urodynamics testing has determined these symptoms result from uninhibited bladder contractions, and so anticholinergic drugs that control these contractions are the mainstay of therapy typically given in six monthintervals until the condition resolves. Beyond the embarrassment that may accompany urinary incontinence, US has been linked to urinary tract infection (UTI) and vesicoureteral reflux. Specifically, among females with UTI, at least 40% also have US, and US has been identified as a cause for reflux and a factor that delays its otherwise expected spontaneous resolution. Consequently, identification and treatment of US are important to the management of children with UTI, reflux and/or incontinence.

Constipation also has been associated with UTI, vesicoureteral reflux, and urinary incontinence in children. Although these observations date at least to the 1950s, relatively few studies have attempted either to establish the incidence of constipation found with these various pediatric urologic conditions, or to document the impact of bowel therapy upon their management. Of these, Yazbeck et al studied 47 children with recurrent UTI and noted all were constipated and had uninhibited bladder contractions during urodynamics testing. Therapy directed toward relief of constipation resolved bladder symptoms in 25%. Loening-Baucke reported 46% of 234 children attending a university-based encopresis clinic also experienced urinary incontinence, which diminished with laxative therapy. A recent evaluation of 582 children with US estimated that 16% were also constipated based upon a history of bowel activity.

We have been concerned about the apparent association between US and constipation, especially since anticholinergic drugs commonly prescribed for uninhibited bladder contractions could exacerbate underlying stool retention and thereby prolong bladder dysfunction. It is also our experience that parents are not very familiar with bowel activity of their children after the usual age of toilet training, making history potentially unreliable for diagnosing constipation. Therefore, we started recommending a brief course of laxatives for all patients presenting with US, reserving anticholinergics for those whose bladder symptoms persisted. In a retrospective review of 110 children, we found 34% had relief of bladder symptoms with laxatives alone, so that anticholinergic medications were not then required, and the history of whether the child was constipated or not did not predict response. However, this study has been criticized for not being placebo-controlled.

Given the potential impact of this observation for the management of children with not only urinary incontinence but also UTI and reflux who have US, we now propose a prospective, randomized, double-blinded, placebo-controlled study of the impact of laxative therapy upon children with US.

ELIGIBILITY:
Inclusion Criteria:

* Toilet-trained with a history of urinary tract infection
* Vesicoureteral reflux
* Urinary incontinence
* Daily frequency and urgency
* Diurnal incontinence.

Exclusion Criteria:

* Children who are below 4 years old as they may still not be toilet-trained;
* Children with encopresis
* Children with anorectal malformations
* Children with neurologic disorders

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2007-12-10 (Actual); Primary Completion 2014-06-17 (Actual); Study Completion 2014-07-22 (Actual)

PRIMARY OUTCOMES:
Mean change in USQ (Urinary Symptom Questionnaire) scores | Baseline,1 month
  Vancouver urinary symptom questionnaire (USQ) measures urinary urge symptom with possible score range from 0 (no urge symptoms) to 16 (all 4 symptoms occurring almost always), with higher ΔUSQ demonstrating greater symptom improvement (i.e. less urinary urge symptoms)
Mean change in BSQ (Bowel Symptom Questionnaire) scores | Baseline, 1 month
  Bowel symptom questionnaire (BSQ) measures bowel symptoms with possible score range from 0-20 with higher ΔBSQ demonstrating greater symptom improvement

SECONDARY OUTCOMES:
Number of patients with constipation | 1 month
  The evidence of constipation was measured by abdominal X-ray (KUB) (kidneys, ureters, and urinary bladder)

CONTACTS AND LOCATIONS:
Overall Officials: Warren T Snodgrass, MD, Principal Investigator — PARC Urology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bush NC, Shah A, Barber T, Yang M, Bernstein I, Snodgrass W. Randomized, double-blind, placebo-controlled trial of polyethylene glycol (MiraLAX(R)) for urinary urge symptoms. J Pediatr Urol. 2013 Oct;9(5):597-604. doi: 10.1016/j.jpurol.2012.10.011. Epub 2012 Nov 3. PMID 23127806